CLINICAL TRIAL: NCT00563927
Title: Prospective Randomized Study on Therapeutic Gain Achieved By Addition of Chemotherapy for T1-4N2-3M0 Nasopharyngeal Carcinoma
Brief Title: Benefit of Adding Chemotherapy for Advance Nasopharyngeal Carcinoma (T1-4N2-3M0)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital Authority, Hong Kong (Other Government)
Collaborators: Hong Kong Nasopharyngeal Cancer Study Group Limited (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: L/M-77 TO PYH08/79; HARECCTR0500023; NPC99-01
Record Dates: First submitted 2007-11-21; First posted 2007-11-26 (Estimated); Last update posted 2010-07-07 (Estimated); Status verified 2010-07

CONDITIONS: Nasopharyngeal Neoplasms; Carcinoma, Squamous Cell
Keywords: Nasopharyngeal Carcinoma; T1-4N2-3M0
MeSH Terms: conditions — Nasopharyngeal Neoplasms; Carcinoma, Squamous Cell; Nasopharyngeal Carcinoma | interventions — Cisplatin; Fluorouracil

INTERVENTIONS:
Procedure: Conventional RT
Drug: Cisplatin
Drug: 5-fluorouracil

SUMMARY:
To test the therapeutic ratio of additional chemotheray on advanced nasopharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Undifferentiated or non-keratinizing carcinoma
* Tumor staged as N2-3
* No evidence of distant metastasis M0
* Performance status:0-2
* Marrow: WBC >= 4 and platelet >= 100
* Renal: creatinine clearance >= 60
* Informed consent

Exclusion Criteria:

* WHO type I squamous cell carcinoma or adenocarcinoma
* Age >= 70
* Palliative intent or tumor extent mandating AP opposing facio-cervical fields
* Prior malignancy except adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease-free for 5 years
* Previous radiotherapy (except non-melanomatous skin cancers outside the intended RT treatment volume
* Previous chemotherapy
* Patient is pregnant or lactating

Max Age: 70 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 1999-03; Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
Failure free survival rate | 5 year

SECONDARY OUTCOMES:
Disease-specific survival rate | 5-year
Overall survival rate | 5-year
Complication-free rates | 5-year

CONTACTS AND LOCATIONS:
Overall Officials: Wai Hon LAU, Dr, Principal Investigator — Department of Clinical Oncology, Queen Elizabeth Hospital
Locations (4):
- China (4):
  - Pamela Youde Nethersole Eastern Hospital, Hong Kong
  - Queen Elizabeth Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
  - Tuen Mun Hospital, Hong Kong